CLINICAL TRIAL: NCT06459921
Title: Efficacy and Safety of Neoadjuvant Sintilimab Puls FLOT Versus Sintilimab Puls SOX Phase II Clinical Trial for Patients With Locally Advanced Gastric Cancer
Brief Title: Efficacy and Safety of Neoadjuvant Sintilimab Plus FLOT Versus Sintilimab Plus SOX Phase II Clinical Trial for Patients With Locally Advanced Gastric Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: loong-201
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-04

CONDITIONS: Neoadjuvant Chemotherapy; Sintilimab; Locally Advanced Gastric Cancer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FLOT+Sintilimab (Active Comparator): Patients in the FLOT group received 4 cycles of standard FLOT chemotherapy, the FLOT chemotherapy cycle consists of: day 1: intravenous 5-FU 2600 mg/m² inserted through a peripherally inserted central catheter (PICC) for 24 hours intravenous folic acid 200 mg/m2 intravenous OXA 85 mg/m² intravenous TXT 50 mg/m². The next cycle of chemotherapy was repeated on day 15. Sintilimab: 200 mg every 3 weeks.
  Interventions: Drug: FLOT+Sintilimab
- SOX+Sintilimab (Experimental): Patients in the SOX group received 3 cycles of S-1 + OXA chemotherapy prior to radical gastrectomy.The SOX chemotherapy cycle consists of: day 1: intravenous OXA 130 mg/m² days 1-14: oral S-1 80 mg/m², 2 times/Day. Repeat next chemotherapy on day 22. Sintilimab: 200 mg every 3 weeks.
  Interventions: Drug: SOX+Sintilimab

INTERVENTIONS:
Drug: SOX+Sintilimab — Patients would be allocated to the SOX+Sintilimab group.
  Arms: SOX+Sintilimab
Drug: FLOT+Sintilimab — Patients would be allocated to the FLOT+Sintilimab group.
  Arms: FLOT+Sintilimab

SUMMARY:
This study aims to investigate the efficacy and safety of Sintilimab combined with FOLT versus Sintilimab combined with SOX in patients with locally advanced gastric cancer. The research design is intended to observe the comparison of conversion therapy effects, disease-free survival, R0 resection rate, and safety evaluation between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age >=18 years and <100 years.
* 2. Diagnosed with locally advanced gastric cancer.
* 3. Eastern Cooperative Oncology Group ECOG PS score 0-1.
* 4. adoption of preoperative chemotherapy treatment and PD-1 antibody therapy.
* 5. deficient mismatch repair identified by pathological detection.

Exclusion Criteria:

* 1. Locally advanced unable to resect or metastatic tumors.
* 2. Patients with recurrence of residual gastric cancer
* 3. Patients refusing surgical resection after preoperative chemotherapy therapy.
* 4. Have received any anti-tumor therapy such as chemotherapy, radiotherapy, immunotherapy, etc., or have been more than 180 days since the last treatment.
* 5. Patients with confirmed allergy to the study drug and/or its excipients.
* 6. Severe malnutrition and active autoimmune diseases.
* 7. Pregnant or lactating women.
* 8. Patients with medical systemic diseases and psychiatric diseases that are not amenable to chemotherapy.
* 9. Patients with acute infections requiring antibiotic treatment.
* 10. Patients with acute infections requiring antibiotic treatment.
* 11. Patients who are concomitantly receiving other immunotherapy, corticosteroids, and other anticancer therapies during the trial.
* 12. Positive test result for hepatitis B or hepatitis C virus.
* 13. Untreated central nervous system metastatic peripheral neuropathy (>grade 1).
* 14. History of malignancy within the past 5 years (with the exception of curative, localized cancer).
* 15. Patients who are not expected to achieve R0 resection.
* 16. Weight loss greater than or equal to 20% within 4 weeks before the first dose.
* 17. Patients with multiple factors affecting oral medication.
* 18. Vaccination within 4 weeks prior to the first dose of study drug.
* 19. Patients who have received immune checkpoint inhibitors and develop serious adverse reactions after treatment and need to be permanently disabled.
* 20. The investigator believes that the subject has other serious systemic diseases or other reasons and is not suitable for this clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of radical (R0) resection after neoadjuvant therapy | From the preoperative chemotherapy until the occurrence of adverse events, assessed up to 180 days
  efficacy of Sintilimab combined with FOLT versus Sintilimab combined with SOX in patients with locally advanced gastric cancer.

SECONDARY OUTCOMES:
adverse event | From the preoperative chemotherapy until the occurrence of adverse events, assessed up to 180 days
  adverse event caused by FLOT, SOX or Sintilimab treatment, which were coded using the Medical Dictionary Regulatory Activities version 20.1 and adverse event grade according to the National Cancer Institute Common Terminology Criteria for Adverse Events
disease-free survival | From date of diagnosis until the first documented recurrence or death, assessed up to 60 months
  from diagnosis to recurrence or death

IPD SHARING:
Plan to Share IPD: No